CLINICAL TRIAL: NCT06193083
Title: DEprescribing: Perceptions of PAtients Living With Advanced Cancer. A Multicentre, Prospective Mixed Observational Study
Brief Title: DEprescribing: Perceptions of PAtients Living With Advanced Cancer
Acronym: DEPAL
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Fondation de France (Other); Nantes University (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC23_0563
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-06

CONDITIONS: Deprescribing; Palliative Care; Oncology
Keywords: Deprescribing; Palliative care; Oncology
MeSH Terms: conditions — Neoplasms | interventions — Functional Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qualitative study: The study will comprise an initial qualitative phase. Semi-directed individual interviews using a descriptive approach will be carried out (around 25 patients, over an 8-month period).
  Interventions: Other: Semi-directed individual interviews
- Quantitative study: Following analysis of the qualitative data, we will then carry out a quantitative study to determine the distribution of the different profiles within this population and the factors influencing the perception of deprescription. The self-administered questionnaires, rPATD and BMQ (medication beliefs questionnaire), potentially supplemented by other items following analysis of the qualitative data, will be administered to 300 patients (over a 12-month period).
  The ancillary study will be carried out during this second phase, using a validated self-questionnaire to assess patients' level of literacy.
  Interventions: Other: The self-administered questionnaires, rPATD and BMQ; Other: The self-administered FCCHL (Functional, Communicative and Critical Health Literacy) / HLS14 (14-item health literacy scale)

INTERVENTIONS:
Other: Semi-directed individual interviews — Individual semi-structured interviews (descriptive approach methodology with reflexive thematic analysis)
  Groups: Qualitative study
Other: The self-administered questionnaires, rPATD and BMQ — rPATD: The rPATD is a questionnaire validated and adapted in French to assess patients' perceptions of their treatments and deprescribing.
  This self-administered questionnaire consists of 22 questions rated on a 5-point Likert scale (scale from 1 to 5, at 1 the patient completely agrees with the questionnaire's proposal, at 5 the patient strongly disagrees with the questionnaire's proposal). Following the analysis of Phase 1 "Qualitative" of the protocol, three additional questions
  BMQ French version of the BMQ self-questionnaire, which studies patients' perceptions of medication .
  The Beliefs about Medicine Questionnaire (BMQ) is an 18-item self-administered questionnaire designed to explore patient perceptions of medicine. It has been validated in French and is free to use.
  It comprises 10 items relating to specific beliefs about prescribed treatments:
  A 5-point Likert-type scale was used for each item. The higher the sum of the scores obtained, the stronger the subject's belief.
  Groups: Quantitative study
Other: The self-administered FCCHL (Functional, Communicative and Critical Health Literacy) / HLS14 (14-item health literacy scale) — FCCHL (Functional, Communicative and Critical Health Literacy)/HLS14 (14-item health literacy scale) (https://reflis.fr/wp-content/uploads/2020/07/FCCHL-HLS14-Questionnaire-Litteratie-sante.pdf )
  Validated French-language self-administered questionnaire and consisting of14 items with a 5-point Likert scale for assessing health literacy :
  Functional literacy: basic reading and writing skills sufficient to function effectively in everyday situations Communicative or interactive literacy: more advanced cognitive and literacy skills that, combined with social skills, can be used to actively participate in everyday activities, extract information and meanings from different forms of communication, and apply new information to changing circumstances Critical literacy: more advanced cognitive skills which, combined with social skills, can be applied to the critical analysis of information and the use of that information to exercise greater control over life events and situations
  Groups: Quantitative study

SUMMARY:
Polymedication in palliative oncology care is a real public health problem. This phenomenon has been shown to increase the risk of iatrogenesis, reduce patients' quality of life and increase healthcare costs. For many years, health policies have been developed in geriatrics to reduce polymedication through deprescription tools.

Recently, palliative care initiatives have been introduced, but without having studied the potential specificities of this population (younger, with a different care dynamic and life trajectory). It is important to better understand this population's perceptions of deprescribing in order to adapt tools/actions to make these approaches more efficient.

The primary aim of this study is to investigate patients' perceptions of deprescribing in palliative cancer care, and the secondary aim is to investigate factors that may influence patients' attitudes and beliefs about deprescribing. At the same time, we will study the psychometric properties of the rPATD (Revised Patients' Attitudes Towards Deprescribing) in this population (a standardized questionnaire validated in geriatric medicine to assess patients' perceptions of deprescription).An ancillary study will be carried out to investigate the link between patients' health literacy and their perception of deprescribing (health literacy is defined as the ability to acquire, understand and use information in ways that promote and maintain good health).

To meet our objectives, we will conduct a 3-year national, prospective, observational, multicenter study with an exploratory sequential mixed design. The study will comprise an initial qualitative phase. Semi-directed individual interviews using a descriptive approach will be carried out (around 25 patients, over an 8-month period). Following analysis of the qualitative data, we will then carry out a quantitative study to determine the distribution of the different profiles within this population and the factors influencing the perception of deprescription. The self-administered questionnaires, rPATD and BMQ (medication beliefs questionnaire), potentially supplemented by other items following analysis of the qualitative data, will be administered to 300 patients (over a 12-month period).The ancillary study will be carried out during this second phase, using a validated self-questionnaire to assess patients' level of literacy.

Thanks to the different results, we will improve our knowledge of the perception of deprescription in palliative oncology care, in order to develop approaches adapted to the specificities of our population to reduce polymedication and thus improve the quality of life of our patients and reduce the risks of iatrogenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Locally advanced or metastatic solid cancer (i.e., palliative care as defined by the World Health Organization)
* Life expectancy estimated by the physician at inclusion of less than 1 year (use of surprise question to help clinician estimate life expectancy)
* Hospitalized or in consultation
* With at least one PIMs (identified using STOPPfrail 2)
* Patient not having expressed opposition to participating in the study after receiving information from the physician.

For qualitative study patients :

- Patients who have signed an authorization for the recording of their voice during the semi-structured interview for the purpose of written transcription.

Exclusion Criteria:

* Minor
* Major under guardianship, protected person
* Patient unable to speak or write French
* Patient with impaired judgment, cognitive or sensory impairment that prevents him/her from receiving informed information, answering questionnaires or participating in a study interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We'll be looking at major patients with "solid" cancer in a palliative situation (locally advanced or metastatic cancer, thus requiring palliative care as defined by the World Health Organization), who have at least one PIMs, followed up on an inpatient or outpatient basis, with a life expectancy estimated at less than 1 year by the doctor caring for the patient.
  To identify whether a patient has at least one PIMs, we will use the STOPPFrail 2 tool . This is a tool developed in geriatrics, validated for a population with an estimated life expectancy of less than 1 year, and which is not specific to oncology. Life expectancy of less than one year will be estimated by the question surprised by the doctor caring for the patient ("Would you be surprised if your patient died within a year?") .
  We will carry out a multicenter study in oncology and/or palliative care departments of hospitals located in western France.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
To study patients' perceptions of deprescribing in palliative cancer care. | at study inclusion
  To describe, understand and explain patients' attitudes and beliefs concerning deprescribing by means of individual semi-structured interviews (descriptive approach methodology with reflexive thematic analysis) and secondly using the rPATD questionnaire (questionnaire for assessing patients' perceptions of their treatments and deprescribing), which can be adapted following analysis of qualitative data.
  rPATD: The rPATD is a questionnaire validated and adapted in French to assess patients' perceptions of their treatments and deprescribing.
  This self-administered questionnaire consists of 22 questions rated on a 5-point Likert scale

SECONDARY OUTCOMES:
To investigate factors that may influence patients' attitudes and beliefs regarding de-prescribing. | at study inclusion
  Influence of gender, age, level of education, type of cancer, number of metastatic sites, Performans status score, presence of systemic cancer treatment (chemotherapy, targeted therapy, immunotherapy, hormonal therapy, etc.), follow-up by a palliative care team, and other factors. ), follow-up by a palliative care team, patient's place of care, persons in charge of treatment, number of medications, number of potentially inappropriate medications (PIMs), prognosis assessed by the referring physician, patient's level of education and beliefs about treatments in general (BMQ questionnaire) on scores from the rPATD questionnaire.
To evaluate the psychometric properties of the rPATD in this population. | at study inclusion
  Description of rPATD validation data in our population: validation of questionnaire structure, measurement of score reliability, concurrent validation with the BMQ questionnaire.
  BMQ French version of the BMQ self-questionnaire, which studies patients' perceptions of medication .
  A 5-point Likert-type scale was used for each item. The higher the sum of the scores obtained, the stronger the subject's belief.

OTHER OUTCOMES:
ANCILLARY STUDY | at study inclusion
  For patients who wish to do so (depending on their fatigability), we will study the link between patients' level of health literacy and their perception of deprescribing (health literacy is defined as the ability to acquire, understand and use information in ways that promote and maintain good health ).
  To do this, we will assess the link between patients' level of literacy (using the FCCHL (Functional, Communicative and Critical Health Literacy) / HLS14 (14-item health literacy scale) self-questionnaire) and their perception of deprescription.

CONTACTS AND LOCATIONS:
Overall Officials: Adrien EVIN, Principal Investigator — Nantes University Hospital
Locations (8):
- France (8):
  - CHD Vendée, La Roche-sur-Yon
  - Hospices Civils de Lyon, Lyon
  - CHU de Nantes, Nantes
  - USP - Maison de Nicodème, Nantes
  - Hôpital Institut CURIE, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CH ST Nazaire, Saint-Nazaire
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evin A, Bourdon M, Nizet P, Hardouin JB, Victorri-Vigneau C, Huon JF. DEprescribing: Perceptions of PAtients living with advanced cancer. A multicentre, prospective mixed observational study protocol. PLoS One. 2024 Aug 20;19(8):e0305737. doi: 10.1371/journal.pone.0305737. eCollection 2024. PMID 39163415